CLINICAL TRIAL: NCT06948812
Title: Effect of Various Initial Foot Positions on Proprioception, Balance, Jump, and Electromyographical Muscle Activity in Basketball Players With Flatfoot and Chronic Ankle Instability: A Cross-sectional Study
Brief Title: Foot Positions Affect Basketball Players With Flatfoot
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Associate Lecturer, Beni-Suef University
Other Study IDs: BNS2
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Balance; Proprioception; Jumping Performance; EMG
Keywords: basket ball players; balance; flatfoot; electromyography; propioception
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- flexible FF: 28 basketball player with flexible flatfoot and chronic ankle instability
- Rigid FF: 28 basketball player with rigid flatfoot and chronic ankle instability
- Control: 28 basketball player without flatfoot but chronic ankle instability

SUMMARY:
This study investigated the effect of various initial foot positions on knee and ankle proprioception, balance, dynamic balance, vertical jump, and electromyographical muscle activity in basketball players with FF.

DETAILED DESCRIPTION:
Objective: To investigate the effect of various initial foot positions on knee and ankle proprioception, balance, dynamic balance, vertical jump, and electromyographical muscle activity in basketball players with FF.

Methods: Eighty-four basketball players with chronic ankle instability were distributed to three groups (28 with flexible FF, 28 with rigid FF, and 28 without FF). The outcome measures will include static and dynamic balance, knee and ankle proprioception, vertical jump, and electromyography (EMG) of ankle muscles (including gastrocnemius (GE), soleus (SOL), tibialis anterior (TA), and peroneus longus (PL) muscles)

ELIGIBILITY:
Inclusion Criteria:

* The presence of flatfoot in the dominant leg.
* The presence of chonic ankle instability

Exclusion Criteria:

* The exclusion criteria were the existence of limited hallux dorsiflexion
* previous hip, pelvis, knee, or foot surgeries within the last year; obesity or pregnancy; leg-length discrepancies;
* Had any vestibular disorder neurological disorder, brain concussion within the last 3 months that may cause balance impairment; or administering any drugs that could disturb alertness or balance

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Basketball players with chronic ankle instability
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Knee proprioception with repositioning error test | 3 months
  The knee proprioception will be measured using the repositioning error test on the dominant leg to measure the absolute angular error. This test will assess the ability of the participant to reproduce a previously performed position (45 and 15 degrees of knee flexion).
Ankle proprioception with angular error measurement test | 3 months
  This test will assess the ability of the participant to reproduce previously performed ankle positions (15° dorsiflexion and 15° plantar flexion.)
Static balance with The Y-Balance test | 3 months
  The Y-Balance test will be used to evaluate static balance 27. The test will assess the ability of the participant to maintain balance while reaching as far as possible in all three directions (anterior (A), posteromedial (PM), and posterolateral (PL) directions).
Dynamic balance with Biodex Balance device | 3 months
  In this study, dynamic balance will be measured by the Biodex Balance System (Biodex 945-302, Biodex Medical Systems Inc., New York, USA). The Biodex Balance System has been demonstrated to be a reliable and validated instrument to assess dynamic balance. The biodex will assess the anteroposterior and lateral stability.
Vertical jump height with vertical jump tester | 3 months
  A vertical jump tester (Sports Imports, Columbus, OH)32 will be utilized to evaluate the vertical jump height in cm of each participant. The achieved height distance in cm in each step will be recorded, and the maximum height will be used in the statistical analysis.
Electromyographical activity (EMG) during one-leg standing | 3 months
  A wireless surface EMG system will record electromyographical signals (EMG) of ankle muscles, including gastrocnemius (GE), soleus (SOL), tibialis anterior (TA), and peroneus longus (PL) muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Nahda University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided